CLINICAL TRIAL: NCT06292117
Title: Implementation of Onsite Rapid CYP2C19 Assay for Genotype Guided Dual Antiplatelet Therapy After Acute Ischemic Stroke
Acronym: ORCA-AIS
Status: Recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Rachael Stone, Principal Investigator, University of Virginia
Other Study IDs: 230247
Record Dates: First submitted 2024-02-25; First posted 2024-03-04 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Ischemic Stroke; CYP2C19 Polymorphism
Keywords: pharmacogenomics; pharmacogenetics; dual antiplatelet therapy; secondary prevention of ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples and extracted DNA from each participant who consents to specimen banking will be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CYP2C19 Genotype — qPCR-based genotyping assay interrogating all Association for Molecular Pathology (AMP) recommended Tier 1 and Tier 2 single nucleotide polymorphisms (SNPs) for CYP2C19 (*2, *3, *4, *5, *6, *7, *8, *9, *10, *17, *35)

SUMMARY:
The goal of this observational study is to use a genetic test to help doctors prescribe the most effective medications after a patient has a stroke. One type of stroke is caused by a blood clot in brain vessels. After a patient has this kind of stroke, they are often given a combination of two blood thinners to prevent it from happening again. One of these blood thinners, called clopidogrel, is less effective in some people due to differences in their DNA. Clopidogrel needs to be activated by a specific enzyme in the body known as CYP2C19. This enzyme does not work as well if there are variations in the section of DNA that tells the body how to make CYP2C19. It can be predicted who has less CYP2C19 enzyme activity with a genetic test. If these patients are given a different blood thinner, it can reduce their risk of another stroke compared to if they are given clopidogrel.

The main questions this study aims to answer are:

* What are the best strategies to implement this genetic test in the hospital?
* Does implementation of this genetic test change providers' decisions on which medication to prescribe after a participant has a stroke?

Participants in this study will have a genetic test done onsite looking for variations in the section of DNA that tells the body how to make CYP2C19. This genetic test will only look for 11 known variations; the genome will not be sequenced. The investigators will alert the doctor of the patient's test results so they can prescribe the appropriate blood thinner. Through this, the investigators will learn the best practices for successful implementation of this genetic test.

DETAILED DESCRIPTION:
Dual antiplatelet therapy (DAPT) with clopidogrel and aspirin is the standard of care (SOC) for secondary prevention of non-cardioembolic minor acute ischemic stroke (AIS) and high-risk transient ischemic attack (TIA); however, clopidogrel has limited effectiveness in CYP2C19 loss-of-function (LOF) allele carriers. Recent studies have demonstrated the superiority of ticagrelor over clopidogrel in CYP2C19 LOF allele carriers, especially when started within 24 hours of presentation. However, despite evidence of improved efficacy and advances in rapid genotyping technology, clinical care has been slow to adopt this form of precision medicine. To address this gap, an implementation study will be conducted in adult patients with cerebrovascular disease to determine the feasibility and acceptability of rapid CYP2C19 genotyping in an acute inpatient setting and to analyze the impact of this clinical implementation on DAPT prescribing patterns. To accomplish these aims, patients undergoing evaluation for AIS/TIA in the Emergency Department will be consented for in-house rapid quantitative polymerase chain reaction (qPCR) genotyping of CYP2C19. Genotype results will be recorded in the electronic health record and active clinical decision support alerts will be built to inform prescribers of any recommended DAPT changes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years of age
* Presenting with symptoms of acute ischemic stroke or transient ischemic attack and without contraindications to dual antiplatelet therapy at time of clinical research coordinator screening
* Presenting within 24 of symptom onset; or, within 24-96 hours of symptom onset IF planned to receive or already on dual antiplatelet therapy

Exclusion Criteria:

* Receiving therapeutic anticoagulation or clear indication for initiation of anticoagulation after event (e.g., known atrial fibrillation)
* History of allogeneic bone marrow transplant
* History of liver transplant
* Subject who is unable to consent and does not have a surrogate available to consent on their behalf

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals evaluated in the Emergency Department or admitted inpatient at an academic medical center
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients discharged from University of Virginia (UVA) Health on dual antiplatelet therapy with a diagnosis of AIS/TIA meeting eligibility criteria upon presentation that are successfully genotyped | At time of participant discharge from hospital; approximately 1-5 days
Average turnaround time of genotype result from time of collection of blood sample to time result is entered into the electronic health record | From time of participant blood draw up to 21 days after

SECONDARY OUTCOMES:
Number of CYP2C19 LOF carriers for whom a genotype-guided modification to DAPT is made | Within 30 days of participant index event
Number needed to genotype (NNG): number of patients who would need to undergo genotyping to have a recommended change in DAPT based on genotype | Within 30 days of participant index event
Stroke-free status via the Questionnaire to Verify Stroke-Free Status (QVSFS) of participants at 90 days in participants who received DAPT | 90 days after participant index event
Major adverse cardiovascular events at 90 days in participants who received DAPT | 90 days after participant index event
Correlation between P2Y12 reaction units (PRUs) measured via P2Y12 assay and CYP2C19 genotype in patients who received DAPT | During participant admission, approximately 1-3 days
  P2Y12 assay collected at least 12 hours after loading dose of P2Y12 inhibitor OR after three doses of maintenance dose if did not receive loading dose

OTHER OUTCOMES:
Acceptability of deferred consent process in participants approached for full informed consent | At time of 90-day follow-up
  Structured interview and/or written survey with pre-specified questions
Cost-effectiveness of CYP2C19-guided dual antiplatelet therapy after acute ischemic stroke | From time of participant blood draw up to 90 days after
  Cost-effectiveness analysis reporting incremental cost-effectiveness ratios (ICER)

CONTACTS AND LOCATIONS:
Overall Officials: Rachael M Stone, PharmD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data may be made available after reasonable request to the PI